CLINICAL TRIAL: NCT05407363
Title: Ridge Augmentation With Simultaneous Implant Placement Using Xenogenic Blocks or Autogenous Bone Blocks With Autogenous Tooth Graft
Brief Title: Ridge Augmentation With Simultaneous Implant Placement Using Bone Blocks With Autogenous Tooth Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, Director, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-72
Record Dates: First submitted 2022-04-01; First posted 2022-06-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Ridge Augmentation; Implant; Autogenous Tooth Graft
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABB and ATG with simultaneous implant placement (Experimental): Using ABB with ATG to fill the gap around simultaneously placed dental implants
  Interventions: Procedure: ABB and ATG with simultaneous implant placement
- XBB and ATG with simultaneous implant placement (Experimental): Using XBB with ATG to fill the gap around simultaneously placed dental implants
  Interventions: Procedure: XBB and ATG with simultaneous implant placement
- ABB and ABG with immediate implant (Active Comparator): Using ABB with ABG to fill the gap around immediately placed dental implants
  Interventions: Procedure: ABB and ABG with simultaneous implant placement

INTERVENTIONS:
Procedure: ABB and ATG with simultaneous implant placement — Ridge augmentation using ABB and ATG as a graft material with simultaneous implant placement
  Arms: ABB and ATG with simultaneous implant placement
Procedure: XBB and ATG with simultaneous implant placement — Ridge augmentation using XBB and ATG as a graft material with simultaneous implant placement
  Arms: XBB and ATG with simultaneous implant placement
Procedure: ABB and ABG with simultaneous implant placement — Ridge augmentation using ABB and ABG as a graft material with simultaneous implant placement
  Arms: ABB and ABG with immediate implant

SUMMARY:
Autogenous bone, with its osteogenic, osteoinductive, and osteo-conductive characteristics has been used for bone grafts with optimal integration into host tissues. For this reason, autogenous bone has been often considered the gold standard of bone regeneration material. However, the amount of autogenous bone that may be harvested is limited, and the harvesting procedure is traumatic.

Bone substitutes, including allografts, xenografts, and alloplasts have been used successfully as alternatives to autogenous bone grafts in ridge augmentation procedures.

In 2008, autogenous tooth bone graft (ATG) was introduced and used for the first time as a bone grafting material for GBR. The tooth contents are extremely similar to that of the alveolar bone. The enamel inorganic, organic, and water contents are 95 percent, 0.6 percent, and 4 percent, respectively. However, in the dentin, the percentages are 70 to 75 percent, 20 percent, and 10 percent, respectively. They are 65 percent, 25 percent, and 10 percent, respectively, when compared to the alveolar bone content.

The aim of this study is to compare ridge augmentation using autogenous bone block (ABB) with immediate implant placement and filling the generated gap with autogenous bone graft (ABG) or ATG, or ridge augmentation using xenograft bone block (XBB) with immediate implant placement and filling the generated gap with ATG.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with buccal bone destruction by periodontal disease and need extraction (horizontal or vertical bone defect);
* Absence of acute inflammation;
* Absence of uncontrolled systemic illness that would preclude implantation;
* Good dental and systemic healthy conditions;
* Patients were willing and able to return for multiple follow-up visits.

Exclusion Criteria:

* Patients with systemic illnesses,
* psychological abnormalities,
* para-functional habit,
* smokers or alcoholics,
* pregnant and lactating patients,
* patients undergoing or recently completed radiotherapy or chemotherapy,
* patients on drugs affecting the healing process,
* patients with endodontically treated teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation probing pocket depth and amount of bone around simultaneously placed dental implants | 9 months
  Changes on pocket depth and amount of bone using ABG or ATG with ABB or XBB around simultaneously placed dental implants
radiographic outcome measuring the amount of bone around simultaneously placed dental implants | 9 months
  the radiographic outcome by measuring the amount of bone by using ATG or ABG on bone formation with ABB or XBB around simultaneously placed dental implants

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt